CLINICAL TRIAL: NCT05775016
Title: Effects of Adding L-BAIBA to Exercising Adult Overweight and Obese Men and Women on Changes in Body Composition, Glucose Control, and Cardiometabolic Risk Factors
Brief Title: Effects of Adding L-BAIBA to Exercising Adult Overweight and Obese Men and Women
Acronym: LBC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to the withdrawal of funding, which made it impossible to continue the study.
Sponsor: Lindenwood University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-23-29
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Obesity; Weight Loss; Weight, Body; Cardiometabolic Syndrome
Keywords: Obesity; Weight Loss; cardiometabolic syndrome
MeSH Terms: conditions — Obesity; Weight Loss; Body Weight; Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study will be conducted using a double-blind, placebo-controlled, parallel group design.
Who Masked: Participant, Investigator
Masking Description: Intervention will be blinded to both participant and investigators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo (Resistant Dextrin) (n=40)
  Interventions: Behavioral: Exercise
- 750 mg/day Mitoburn (L-BAIBA) (Experimental): 750 mg/day Mitoburn (L-BAIBA)
  Interventions: Behavioral: Exercise
- 1,500 mg/day Mitoburn (L-BAIBA) (Experimental): 1,500 mg/day Mitoburn (L-BAIBA)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 12 week resistance and cardiovascular exercise program

SUMMARY:
Beta-amino isobutyric acid (BAIBA) is a myokine produced in skeletal muscle and has been shown to impact how our body metabolizes fuel. We seek to examine changes in body composition, weight loss, glucose control, and cardiometabolic risk factors after adding supplementation of BAIBA to exercise in overweight and obese men and women.

DETAILED DESCRIPTION:
This study will be conducted using a double-blind, placebo-controlled, parallel group design. Eligible study participants will be randomly assigned to one of three supplementation groups: placebo (resistant dextrin) supplementation + exercise group, 750 mg BAIBA supplementation + exercise group, and a 1500 mg BAIBA supplementation + exercise group. After signing an IRB-approved consent form, prospective participants will be scheduled for a screening visit where they will have their eligibility finalized through completion of a peak VO2 assessment using a motorized treadmill and metabolic cart. Eligible participants will then be fully explained the study and scheduled for a baseline testing session (week 0). Prior to scheduling this visit, participants must complete a 4-day food record. Once a food record is completed, participants will observe an overnight fast and be scheduled to complete the testing session between the hours of 0600 - 1000 hours. Upon arrival, changes in medical status, medications, and dietary supplements will be confirmed before having their body mass and hemodynamics assessed. Next, participants will have their waist circumference, body water (BIS), and body composition (DEXA) assessed to evaluate changes in body composition and obesity status throughout the study protocol. Participants will then have a venous blood sample collected for evaluation of health markers (complete blood counts, comprehensive metabolic panels, and lipid panels) before completing a resting metabolic rate measurement. The resting metabolic rate measurement will be used to prescribe energy intake throughout the study protocol. Participants will then use an electronic tablet and complete the Profile of Mood States and visual analog scales to evaluate perceptions of hunger and appetite. Participants will then be given their first daily dose. All participants will be given instructions and meal plans as well as be offered weekly educational sessions on how to restrict calories and meet protein goals throughout the study protocol. Participants will complete five days per week of exercise consisting of a mixture of walking and resistance training. Daily compliance to the exercise and supplementation groups will be monitored weekly for a 12-week period. Participants who complete at least 80% of their assigned workouts will be considered compliant and will be scheduled for follow-up visits after 6 and 12 weeks of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are between 18 - 60 years of age
* Body mass index values will range from >25.0 to < 32.0 kg/m2, making them qualified as an overweight-to-obese population (https://www.nhlbi.nih.gov/health/educational/lose_wt/BMI/bmicalc.htm)
* Average body mass index for entire study cohort will be less than 30.0 kg/m2. As such an ongoing calculation of the recruited cohort's mean body mass index will be maintained and people will only be randomized into the study if the average cohort body mass index value does not exceed 30.0 kg/m2
* Free-living/uninhibited with use of ambulatory assistive devices (e.g. canes, crutches, walkers, etc.) and independent
* In good health absent of being overweight or mildly obese with no other signs or symptoms of cardiovascular, respiratory, metabolic, immune, psychiatric, or musculoskeletal disease or disorders
* Willingness to maintain consistent sleep duration the evening before study visits
* Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, and carry out all study-related procedures
* Able to complete a peak oxygen consumption exercise test with no contraindications to perform exercise per standards put forth by the American College of Sports Medicine. In other words, they are able to safety complete maximal exercise.

Exclusion Criteria:

* Positive medical history and/or is currently being treated for some form of heart disease, cardiovascular disease
* Currently being treated for kidney disease, renal failure, or has dialysis performed on regular intervals
* Has liver disease or some form of clinically diagnosed hepatic impairment
* Diagnosed with having Type I or Type II diabetes (determined as fasting blood glucose > 126 mg/dL)
* Diagnosed with or is being treated for some form of thyroid disease
* Diagnosed with major affective disorder or other psychiatric disorder that required hospitalization in the prior year
* Diagnosed with some form of immune disorder (i.e., HIV/AIDS)
* History of cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening visit).
* Participant has an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea)
* Positive medical history for any neurological condition or neurological disease
* Currently prescribed a statin drugs (i.e., Lipitor, Livalo, Crestor, Zocor, etc.) or any hypertension medications (i.e., Beta-blockers, ACE Inhibitors, Alpha blockers, Vasodilators, etc.)
* Current smoker (average of > 1 pack per day within the past 3 months) has quit within the past six months. This includes all forms of nicotine
* Intake of any drugs (prescribed or over the counter) or dietary supplements that are known or are purported to weight loss such as thermogenics, hydroxycitric acid, ephedra, capsaicin, etc.
* Participants who are lactating, pregnant or planning to become pregnant
* Have a known sensitivity or allergy to any of the study products
* History of alcohol or substance abuse in the 12 months prior to screening
* Receipt or use of an investigational product in another research study within 30 days of beginning the study protocol
* They plan major changes in lifestyle (i.e., diet, dieting, exercise level, travel, etc.) during the study
* Recent history (<3 months) of exercise training or weight loss (> 5%)
* Any orthopedic limitation that would prevent participation in a general fitness program
* Any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Fat Mass (4-compartment) | 12 weeks
  Changes in Fat Mass (4-compartment)

SECONDARY OUTCOMES:
4-Compartment Lean mass | 12 weeks
  Changes in Lean Mass (4-compartment)
Waist circumference | 12 weeks
  Changes in Waist circumference
Visceral Fat (DEXA) | 12 weeks
  Changes in Visceral Fat (DEXA)
Lean:Fat Ratio (DEXA) | 12 weeks
  Changes in Lean:Fat Ratio (DEXA)
Body Mass | 12 weeks
  Changes in Body Mass
Hunger and appetite visual analog scale | 12 weeks
  Changes in Hunger and appetite visual analog scale
Profile of mood states (POMS) | 12 weeks
  Changes in Profile of mood states (POMS)
Inflammatory markers (e.g. CRP, IL-6, etc.) | 12 weeks
  Changes in Inflammatory markers (e.g. CRP, IL-6, etc.)
Comprehensive Metabolic Panel | 12 weeks
  Changes in Comprehensive Metabolic Panel
Lipid Panel | 12 weeks
  Changes in Lipid Panel
Self-reported adverse events | 12 weeks
  Occurrences of Self-reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Chad M Kerksick, PhD, Principal Investigator — Lindenwood University
Locations (1):
- Exercise and Performance Nutrition Laboratory, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No